CLINICAL TRIAL: NCT06716762
Title: Open vs. Laparoscopic Surgery for Pediatric Choledochal Cyst: A Retrospective Study
Brief Title: Open vs. Laparoscopic Surgery for Pediatric Choledochal Cyst
Status: Completed | Type: Observational
Sponsor: In-Jin Jang (Other)
Collaborators: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Sponsor-Investigator, In-Jin Jang, Professor, Hansung University
Organization: Hansung University (Other)
Other Study IDs: KY20241121
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Congenital Choledochal Cyst; Pediatric Surgery; Surgical Outcomes; Open Surgery; Laparoscopic Surgery
Keywords: Congenital Choledochal Cys; Network Meta-analysis; Robotic-assisted Surgery; Laparoscopic Surgery; Pediatric Surgical Outcomes
MeSH Terms: conditions — Choledochal Cyst | interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open Surgery Group, OSG: This group consists of pediatric patients diagnosed with congenital choledochal cyst (CCC) who underwent open surgery, which involved open cyst excision and Roux-en-Y hepaticojejunostomy. A total of 60 patients were assigned to this group.
  Interventions: Procedure: Open Surgery
- Laparoscopic Surgery Group, LSG: This group includes pediatric patients diagnosed with CCC who underwent laparoscopic surgery, which involved laparoscopic cyst excision and Roux-en-Y hepaticojejunostomy. A total of 12 patients were assigned to this group.
  Interventions: Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Open Surgery — Open cyst excision and Roux-en-Y hepaticojejunostomy performed through a 10 cm incision
  Groups: Open Surgery Group, OSG
Procedure: Laparoscopic Surgery — Laparoscopic cyst excision and Roux-en-Y hepaticojejunostomy performed through small incisions with a laparoscope
  Groups: Laparoscopic Surgery Group, LSG

SUMMARY:
This is a retrospective cohort study designed to compare the outcomes of open surgery versus laparoscopic surgery in pediatric patients diagnosed with congenital choledochal cyst (CCC). The study includes children who underwent surgery at Guangdong Medical University Affiliated Hospital and Guangzhou Women and Children's Medical Center between January 1, 2010, and September 1, 2024. The aim of this study is to evaluate and compare the surgical outcomes, including surgery duration, intraoperative blood loss, hospital stay, and postoperative complications (e.g., bile leakage and intestinal obstruction), between the two surgical approaches. The data collected from the patient records will be analyzed to identify factors influencing surgical outcomes and to guide future treatment decisions for CCC in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients diagnosed with congenital choledochal cyst based on preoperative imaging (e.g., ultrasound, computed tomography（CT）, or magnetic resonance cholangiopancreatography（MRCP)）.

Patients who underwent either open surgery (open cyst excision and Roux-en-Y hepaticojejunostomy) or laparoscopic surgery (laparoscopic cyst excision and Roux-en-Y hepaticojejunostomy) for the treatment of congenital choledochal cyst.

Informed consent for follow-up obtained from the patient's family or legal guardian.

Exclusion Criteria:

Patients lacking one or more key outcome measures, including surgery duration, hospital stay, intraoperative blood loss, incidence of postoperative bile leakage, or incidence of postoperative intestinal obstruction.

Patients with incomplete clinical data, such as missing sex, age, or other essential demographic information.

Patients with coagulation disorders that may interfere with surgery or recovery.

Patients with severe comorbidities or immune system disorders that may complicate surgical intervention or recovery.

Patients who underwent non-surgical treatment (e.g., endoscopic procedures) for congenital choledochal cyst.

Pregnant patients or those who are breastfeeding (if applicable to your study population).

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of pediatric patients diagnosed with congenital choledochal cyst (CCC) who underwent surgical treatment at Guangdong Medical University Affiliated Hospital and Guangzhou Women and Children's Medical Center between January 1, 2010, and September 1, 2024. The total number of patients included in this study is 72, with 60 patients assigned to the open surgery group (OSG) and 12 patients assigned to the laparoscopic surgery group (LSG).
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Surgery Duration | Measured intraoperatively, from the initial incision to the closure of the surgical site, at the end of the surgery.
  The time required to complete the surgical procedure, from the initial incision to the closure of the surgical site. This is measured in minutes and compared between the open surgery and laparoscopic surgery groups
Postoperative Complications | 30 days post-surgery (for short-term complications)
  The occurrence of postoperative complications, specifically bile leakage and intestinal obstruction, in patients undergoing either open or laparoscopic surgery. This is measured as a binary outcome (yes/no) and will be compared between the two groups.
Intraoperative Blood Loss | Measured intraoperatively, during the surgery, from the initial incision to the closure of the surgical site.
  The total amount of blood lost during the surgical procedure, measured in milliliters (mL). This will be compared between the two surgical groups (open surgery and laparoscopic surgery).
Hospital Stay | Measured from the day of surgery to discharge, assessed over the duration of hospital stay, up to 30 days post-surgery.
  The total number of days the patient stays in the hospital post-surgery until discharge. This is compared between the open surgery and laparoscopic surgery groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Hansung University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided